CLINICAL TRIAL: NCT06096675
Title: Pilot Study Evaluating Supervised Cardiac Rehabilitation in Patients With Cardiac Amyloidosis
Brief Title: CAPACITY (Cardiac Amyloidosis and Physical ACtivITY) Study
Acronym: CAPACITY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00095189
Record Dates: First submitted 2023-10-17; First posted 2023-10-24 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Cardiac Amyloidosis
Keywords: heart failure; preserved ejection fraction; cardiac rehabilitation
MeSH Terms: conditions — Amyloid Neuropathies, Familial; Heart Failure | interventions — Cardiac Rehabilitation

STUDY DESIGN:
Intervention Model Description: Enrollment in supervised cardiac rehabilitation for 3 one-hour sessions a week for a total of 12 weeks (36 sessions)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cardiac rehabilitation group (Experimental): Intervention group will have baseline 6-minute walk test and cardiopulmonary exercise test (CPET) testing followed by supervised cardiac rehabilitation program including planned 3 one hour sessions a week for a total of 12 weeks (planned 36 sessions). A post intervention 6-minute walk test and CPET test will be performed within 2 weeks of completion of the 12 week program.
  Interventions: Behavioral: • Cardiac Rehabilitation
- control group - no intervention (No Intervention): Control Group will have baseline 6-minute walk test and CPET testing followed by a repeat 6-minute walk test and CPET test in 12-14 weeks

INTERVENTIONS:
Behavioral: • Cardiac Rehabilitation — Intervention group will have baseline 6-minute walk test and cardiopulmonary exercise test (CPET) testing followed by supervised cardiac rehabilitation program including planned 3 one hour sessions a week for a total of 12 weeks (planned 36 sessions). A post intervention 6-minute walk test and CPET test will be performed within 2 weeks of completion of the 12 week program.
  Other Names: supervised cardiac rehabilitation sessions
  Arms: cardiac rehabilitation group

SUMMARY:
Exercise training in patients with heart failure and preserved ejection fraction (HFpEF) has been associated with an improvement in cardiorespiratory fitness and quality of life.

DETAILED DESCRIPTION:
The Atrium Health cardiac rehabilitation program delivers a comprehensive approach to improve cardiac performance including supervised exercise programs and has the ideal infrastructure to offer cardio-oncology rehabilitation (CORE) to all our cancer patients in the future. Currently neither CORE nor cardiac rehabilitation for HFpEF are covered by insurance, and hence the targeting of a higher risk cancer and non-cancer population of cardiac amyloidosis patients to objectively measure the benefits of a supervised exercise program ultimately to expand eligibility to all cancer patients and shape the treatment and payor landscape in the future.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* New York Heart Association (NYHA) Class I-III Heart Failure
* Able to Exercise
* On stable treatment for their cardiac amyloidosis or under active surveillance
* Life expectancy of at least 6 months
* Ability to understand and the willingness to sign a written informed consent document in English, and the willingness/ability to comply with the protocol activities
* Participant must be able and willing to follow the cardiac rehabilitation activities

Exclusion Criteria:

* Inability to provide informed consent
* Inability to commit to in-person supervised exercise sessions for three one-hour sessions a week for 12 weeks
* NYHA Class IV Heart Failure
* Pulmonary disease requiring home oxygen
* Gait instability or history of prior falls
* In the opinion of the Principal Investigator, have a clinically significant comorbid disease that is likely to affect the ability of the patient to complete the trial, interfere with their ability with measurement of self-reported outcomes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-01-22 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Number of participants that complete at least 75% of prescribed cardiac rehab sessions | Week 12
  Feasibility of cardiac rehab as measured by number of participants that complete at least 75% of prescribed cardiac rehab sessions.

SECONDARY OUTCOMES:
Change in cardiorespiratory fitness - maximal VO2 rates | Week 12
  Change in cardiorespiratory fitness as assessed by maximal (max) rate (V) of oxygen (O₂) your body is able to use during exercise VO2 (ml/kg/min ) on cardiopulmonary exercise test (CPET).
  Vo2 Max scores can vary based on a number of factors in addition to fitness, such as your gender, age and genetics, but a vo2 max measurement for an average person in their mid 30s to mid 40s is likely to be around: Women - 31 ml oxygen/kg of body weight/minute. Men - 42 ml oxygen/kg of body weight/minute.
Change in cardiorespiratory fitness - Ventilatory Efficiency (VE/VCO2) rates | Week 12
  Ventilatory equivalent for carbon dioxide ( ˙VE/ ˙VCO2) identifies the second ventilatory threshold, namely, the point in time when ventilatory drive starts increasing relative to ˙VCO2 (i.e., when hyperventilation occurs).
Change in cardiorespiratory fitness - quality of life (KCCQ) Cardiomyopathy Questionnaire (Kansas City) scores | Week 12
  KCCQ scores are scaled from 0 to 100 and frequently summarized in 25-point ranges, where scores represent health status as follows: 0 to 24: very poor to poor; 25 to 49: poor to fair; 50 to 74: fair to good; and 75 to 100: good to excellent.
Change in cardiorespiratory fitness - chronotropic incompetence scores | Week 12
  the inability of the heart to increase its rate commensurate with increased activity or demand, is common in patients with cardiovascular disease, produces exercise intolerance which impairs quality-of-life - chronotropic incompetence is usually defined as failure to achieve a chronotropic index of 0.8 or higher (i.e., falling below 97.5 percent of healthy adults).
Change in cardiorespiratory fitness - 6-minute walk test distance | Week 12
  In healthy subjects, the 6-min walk distance (6MWD) ranges from 400 to 700 m, the main predictor variables being gender, age and height.

CONTACTS AND LOCATIONS:
Overall Officials: Jai Singh, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Sanger Heart and Vascular Institute, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No